CLINICAL TRIAL: NCT03893903
Title: AMPLIFYing NEOepitope-specific VACcine Responses in Progressive Diffuse Glioma - a Randomized, Open Label, 3 Arm Multicenter Phase I Trial to Assess Safety, Tolerability and Immunogenicity of IDH1R132H-specific Peptide Vaccine in Combination with Checkpoint Inhibitor Avelumab
Brief Title: AMPLIFYing NEOepitope-specific VACcine Responses in Progressive Diffuse Glioma
Acronym: AMPLIFY-NEOVAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT-2016-0458; 2017-000587-15 (EudraCT Number); NOA-21 (Other: Neurooncology Working Group of the German Cancer Society (NOA))
Record Dates: First submitted 2018-08-16; First posted 2019-03-28 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Malignant Glioma
MeSH Terms: conditions — Glioma | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- IDH1 peptide vaccine (Experimental): IDH1R132H peptide vaccine alone
  Interventions: Drug: IDH1R132H peptide vaccine
- combination (Experimental): IDH1R132H peptide vaccine and Avelumab
  Interventions: Drug: IDH1R132H peptide vaccine; Drug: Avelumab
- Avelumab (Experimental): Avelumab alone
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: IDH1R132H peptide vaccine — The vaccine is applied by s.c. injection with 300 μg IDH1R132H peptide emulsified in 0.5 ml 33% DMSO / 0.5 ml Montanide® per dose.
  Patients receive 3 doses in two week intervals for 6 weeks, followed by re-resection. 4 weeks after surgery, treatment will be resumed consisting of 5 additional vaccinations in 4 week intervals, followed by maintenance vaccines until progression in three months intervals after a pause of 16 weeks.
  Arms: IDH1 peptide vaccine; combination
Drug: Avelumab — Avelumab is a humanized anti-PD-L1 antibody approved for patients with Merkel cell carcinoma and urothelial cancer. It is applied by i.v. infusion with 10 mg/kg per dose.
  Patients receive 3 doses of Avelumab in 2week intervals for 6 weeks, followed by re-resection. Avelumab will be administered in monthly intervals starting 4 weeks after the surgery until progression.
  Arms: Avelumab; combination

SUMMARY:
The trial will address safety and tolerability of the combination of the IDH1R132H-specific vaccine with checkpoint blockade and seeks to explore predictive biomarkers for response to checkpoint blockade in post-treatment tumor tissue. The study will enroll 48 evaluable patients (presumably, 60 in total) with IDH1R132H-mutated gliomas with an unfavorable molecular profile (no 1p/19q co-deletion, nuclear ATRX- loss) progressive after radiotherapy and alkylating chemotherapy eligible for re-resection. After diagnosis of recurrent disease on imaging patients will be randomized assigned in a 1:1:2 ratio into three arms. Arm 1 (12 patients) will receive three IDH1R132H peptide vaccines alone in two week intervals. Arm 2 (12 patients) will receive three IDH1R132H peptide vaccines in combination with three doses of Avelumab in two week intervals. Arm 3 (24 patients) will receive three doses of Avelumab in two week intervals. After 6 weeks of treatment patients (Arms 1-3) will undergo planned re-resection. Four weeks after the operation treatment will be resumed consisting of five additional vaccines (Arm 1+2) in 4 week intervals, followed by maintenance vaccines until progression in three months' intervals after a pause of 16 weeks. Avelumab will be administered in monthly intervals in Arms 2 and 3 starting four weeks after the operation until progression.

Key outcome parameters will be safety and immunogenicity (Arms 1 and 2) based on peripheral and intratumoral immune analyses assessed 9 months after re-resection.

DETAILED DESCRIPTION:
The standard of care (SOC) treatment of patients with malignant gliomas is - independent of molecular markers - still confined to surgery, irradiation and alkylating chemotherapy as targeted therapies to date have failed to prove superiority over standard of care in controlled trials. At the same time, novel concepts in immunotherapy have evolved with the identification of potential (neo)epitopes and phase III clinical trials investigating the efficacy of checkpoint inhibitors. Despite patients frequently undergoing resection of recurrent tumor, patient selection criteria for innovative immunotherapy in glioma have been hampered by the lack of availability of post-treatment tumor tissue. Neoepitope-specific vaccines have gained considerable interest also in a challenging disease such as glioma. IDH1R132H, a frequent driver mutation in gliomas, was previously identified to contain a neoepitope. A peptide vaccine targeting this epitope is currently tested in a phase I first-in-man multicenter clinical trial. The clinical phase of this trial was completed in Q3 2017 with 32 patients treated. The primary endpoints were met by demonstrating safety and immunogenicity. Checkpoint inhibitors are tested in unselected populations of glioma patients despite evidence that response is associated with high mutational load, which is infrequent in untreated gliomas, but may occur particularly after long periods of exposure to alkylating chemotherapy.

The trial will address safety and tolerability of the combination of the IDH1R132H-specific vaccine with checkpoint blockade and seeks to explore predictive biomarkers for response to checkpoint blockade in post-treatment tumor tissue. The study will enroll 48 evaluable patients (presumably, 60 in total) with IDH1R132H-mutated gliomas with an unfavorable molecular profile (no 1p/19q co-deletion, nuclear ATRX loss) progressive after radiotherapy and alkylating chemotherapy eligible for re-resection. After diagnosis of recurrent disease on imaging patients will be randomized assigned in a 1:1:2 ratio into three arms. Arm 1 (12 patients) will receive three IDH1R132H peptide vaccines alone in two week intervals. Arm 2 (12 patients) will receive three IDH1R132H peptide vaccines in combination with three doses of Avelumab, a humanized anti-PD-L1 antibody approved for patients with Merkel cell carcinoma and urothelial cancer, in two week intervals. Arm 3 (24 patients) will receive three doses of Avelumab in two week intervals. After 6 weeks of treatment patients (Arms 1-3) will undergo planned re-resection. A safety MRI will be performed three weeks after initiation of the experimental treatment. Four weeks after the operation treatment will be resumed consisting of five additional vaccines (Arm 1+2) in 4 week intervals, followed by maintenance vaccines until progression in three months' intervals after a pause of 16 weeks. Avelumab will be administered in monthly intervals in Arms 2 and 3 starting four weeks after the operation until progression.

Key outcome parameters will be safety and immunogenicity (Arms 1 and 2) based on peripheral and intratumoral immune analyses assessed 9 months after re-resection. Additional exploratory analyses will determine efficacy (all Arms), dependent on predictive molecular immune and imaging biomarkers, such as increased mutational load (Arm 3). Based on the experience in the NOA-04 and CATNON trials the expected time to second progression is 9-12 months.

The trial is supported by the German Cancer Consortium (DKTK) and the Neurooncology Working Group of the German Cancer Society (NOA).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, smoking or non-smoking, of any ethnic origin and gender
* Patients present with unequivocal first, second or third recurrence of a histologically confirmed IDH1R132H-mutated glioma WHO grade II, III or IV progressive after radiotherapy and chemotherapy
* Absence of chromosomal 1p/19q co-deletion in the primary tumor tissue and/or
* Loss of nuclear ATRX expression in the primary tumor tissue (partial loss allowed)
* Availability of tumor tissue for analysis (FFPE bulk tissue)
* Patients have received radiotherapy (54 - 60 Gy) and at least six months of alkylating chemotherapy
* Patients are at least three months off radiotherapy
* Patients must be candidates for re-resection and the re-resection must be postponable for seven weeks
* Patients should be immunocompetent (i.e. no concomitant treatment with dexamethasone (or equivalent), or receive stable/decreasing steroid levels not exceeding 2 mg/day dexamethasone (or equivalent) during the last 3 days prior to clinical screening; no severe lymphopenia)
* Karnofsky Performance Status ≥ 70
* Estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method)
* Ability of patient to understand character and individual consequences of the clinical trial
* Evidence of informed consent document personally signed and dated by the patient (or a witness in case the patient is unable to write) and indicating that the patient has been informed of all pertinent aspects of the study and that the patient consents to participate in the trial
* Women of child-bearing potential (WOCBP; i.e. those who have not undergone a hysterectomy, bilateral salpingectomy and bilateral oophorectomy or who have not been post-menopausal for at least 24 consecutive months) must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of the investigational medicinal product(s) (IMPs).
* WOCBP must be using an effective method of birth control to avoid pregnancy throughout the study and for 3 months after the last dose of the IMP. This includes two different forms of effective contraception (e.g. hormonal contraceptive and condom, IUD/IUS and condom) or sterilization, resulting in a failure rate less than 1% per year.
* Men must be willing and able to use an effective method of birth control throughout the study for up to 3 months after the last dose of the IMP(s), if their sexual partners are WOCBP (acceptable methods see above).
* Availability of pre-study MRT (magnetic resonance tomography) of latest tumor recurrence
* Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Current use of immunosuppressive medication, EXCEPT for the following:

  1. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection);
  2. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent;
  3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Pregnancy or lactation
* Previous or concurrent experimental treatment for the tumor other than radiotherapy and alkylating chemotherapy. This includes local therapies such as interstitial radiotherapy or local chemotherapy (i.e. BCNU wafers), loco-regional hyperthermia, electric fields, and antiangiogenic therapy (such as Bevacizumab).
* Abnormal (≥ Grade 2 CTCAE v4.03) laboratory values for thyroid gland: free T4 and TSH
* Abnormal (≥ Grade 2 CTCAE v4.03) laboratory values for hematology, liver and renal function (serum creatinine). In detail, the following values apply as exclusion criteria:

  1. Hemoglobin < 9 g/dL (5.59 mmol/L)
  2. White blood cell count (WBC) decrease (<3.0 x 109/L) or increase (> 10.0 x 109/L)
  3. Absolute neutrophil count (ANC) decrease (< 1.5 x 109/L)
  4. Platelet count decrease (< 100 x 109/L)
  5. Bilirubin > 1.5 x ULN (upper limit of normal according to the performing lab´s reference range)
  6. ALT > 2,5 x ULN
  7. AST > 2,5 x ULN
  8. GGT > 2.5 x ULN
  9. Serum creatinine increase (> 1.5 x ULN)
* Patients with history or presence of HIV and/or HBV/HCV positivity (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)
* Patients with history or known presence of tuberculosis (positive QuantiFERON®-TB Gold test (or equivalent) or tuberculin skin test). Patients with an indeterminate result of the QuantiFERON®-TB Gold test (or equivalent) are not eligible unless additional testing demonstrates a negative result (tuberculin skin test or repeated QuantiFERON®-TB Gold test/or equivalent). If a tuberculin skin test is performed, an induration of > 6 mm is "positive" for a patient with history of BCG vaccine, while an induration of > 10 mm is "positive" for a patient without history of BCG vaccine. If necessary, a QuantiFERON®-TB Gold or equivalent test might be complemented by additional specific diagnostic tests as per standard procedures.
* Patients with severe infection(s) or signs/symptoms of infection within 2 weeks prior to the first administration of the study drug(s)
* Active infection requiring systemic therapy
* Patients who have received a live, attenuated vaccine within 4 weeks prior to the first administration of the study drug(s)
* Patients with a prior solid organ transplantation or haematopoietic stem cell transplantation
* Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
* Clinically significant (i.e., active) cardiovascular disease: Cerebral vascular accident/stroke (< 6 months prior to enrolment), myocardial infarction (< 6 months prior to enrolment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Persisting toxicity related to prior therapy (NCI CTCAE v.4.03 Grade >1); however, alopecia, sensory neuropathy Grade ≤ 2, or other persisting toxicities Grade ≤ 2 not constituting a safety risk based on investigator´s judgement is acceptable.
* Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3).
* Participation in other clinical trials or their observation period during the last 30 days before the first administration of the IMP(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
safety and tolerability: Regime Limiting Toxicity | Primary treatment phase (week 43)
  To determine safety and tolerability of repeated fixed dose vaccinations of the IDH1 peptide vaccine administered with topical imiquimod (Aldara®) alone (Arm 1) or in combination with Avelumab (Arm 2), or Avelumab alone (Arm 3).
  Primary endpoint is the Regime Limiting Toxicity (RLT) until End of Primary Treatment Phase.

SECONDARY OUTCOMES:
immunogenicity of the IDH1 peptide vaccine | End of primary treatment phase (week 43)
  To assess immunogenicity of the IDH1 peptide vaccine alone or in combination with Avelumab. The main immunogenicity endpoint is the presence of IDH1R132H-specific T-cells and/or antibody responses in the peripheral circulation and/or the presence of IDH1R132H-specific T-cells in the tumor tissue
Frequency of Treatment-Emergent Adverse Events (Assessment of Tolerability) | Time from baseline until EOS (end of study) (12 weeks after last treatment administration); up to 38 months
  This endpoint includes all AEs (adverse event), their severity, SAEs (serious adverse event), the relation of AEs to the study treatment, dose modifications for toxicity and discontinuation of study treatment during the trial phase. Toxic effects will be graded according to CTCAE, current version.
Objective response rate (ORR) to assess the efficacy of Avelumab in association with the number of non-synonymous mutations in the tumor tissue. | Time from baseline until end of the primary treatment phase (week 43) and at EOS (12 weeks after last treatment administration); up to 38 months
  The ORR, defined as the proportion of patients with a treatment-induced hypermutator phenotype compared with a non-hypermutator phenotype showing complete response (CR), partial response (PR) or stable disease (SD) at end of the Primary Treatment Phase and at EOS compared to the baseline value (MRI at visit 7). ORR analysis will be based on the central disease assessment according to the iRANO criteria
Overall survival (OS) | Time from the first study treatment date until death or end of observation (up to 38 months)
  OS, defined as the time from the first study treatment date until death. For patients who do not die, time to death will be censored at the time of the end of observation. The end of observation is defined as the date of study termination as indicated by the corresponding entry of the CRF (case report form). If this date is not documented, the end of observation is defined as the last documented date.
Progression-free survival (PFS) | Time from the day of first study treatment date, censored by the end of the observation (up to 38 months)
  The PFS, defined as time from the day of first study treatment date to the day of tumor progression or the day of death of any cause (whichever occurs first), censored by the end of the observation. The end of observation is defined as the date of study termination as indicated by the corresponding entry of the CRF. If this date is not documented, the end of observation is defined as the last documented date.
Objective response rate (ORR) | Time from baseline until end of the primary treatment phase (week 43) and at EOS (12 weeks after last treatment administration); up to 38 months
  The ORR, defined as the proportion of patients showing complete response (CR), partial response (PR) or stable disease (SD) at end of the Primary Treatment Phase and at EOS compared to the baseline value (MRI at visit 7). ORR analysis will be based on the central disease assessment according to the iRANO criteria
Association between immunogenicity and Objective response rate (ORR) | Time from baseline until EOS (12 weeks after last treatment administration); up to 38 months
  To analyse the association between immunogenicity and the clinical outcome parameter. The clinical outcome will be evaluated by assessing the ORR. Logistic regression models will be used to explore the relationship between the relative changes in the immunologic parameters and ORR.
Association between immunogenicity and Progression-free Survival (PFS) | Time from baseline until EOS (12 weeks after last treatment administration); up to 38 months
  To analyse the association between immunogenicity and the clinical outcome parameter. The clinical outcome will be evaluated by assessing the PFS. Proportional Hazards models will be used to analyze the prognostic influence of relative changes in the immunologic parameters, for the PFS.
Association between immunogenicity and Overall survival (OS) | Time from baseline until EOS (12 weeks after last treatment administration); up to 38 months
  To analyse the association between immunogenicity and the clinical outcome parameters. The clinical outcome will be evaluated by assessing the OS. Proportional Hazards models will be used to analyze the prognostic influence of relative changes in the immunologic parameters, for the OS.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Platten, Prof. MD, Principal Investigator — German Canecr Research Center, Heidelberg, and Mannheim University Hospital, Neurology, Mannheim
Locations (10):
- Germany (10):
  - Charité Berlin, Neurosurgery, Berlin
  - University Hospital Dresden, Neurosurgery, Dresden
  - Essen University Hospital, Neurooncology, Essen
  - University Hospital Frankfurt, Neurooncology, Frankfurt am Main
  - University Hospital Freiburg, Neurosurgery, Freiburg im Breisgau
  - University Hospital Heidelberg, Neurology Clinic, Heidelberg
  - Mannheim University Hospital, Mannheim
  - LMU, University Hospital Munich, Munich
  - Katharinenhospital Stuttgart, Neurosurgery, Stuttgart
  - University Hospital Tuebingen, Neurooncology, Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bunse L, Rupp AK, Poschke I, Bunse T, Lindner K, Wick A, Blobner J, Misch M, Tabatabai G, Glas M, Schnell O, Gempt J, Denk M, Reifenberger G, Bendszus M, Wuchter P, Steinbach JP, Wick W, Platten M. AMPLIFY-NEOVAC: a randomized, 3-arm multicenter phase I trial to assess safety, tolerability and immunogenicity of IDH1-vac combined with an immune checkpoint inhibitor targeting programmed death-ligand 1 in isocitrate dehydrogenase 1 mutant gliomas. Neurol Res Pract. 2022 May 23;4(1):20. doi: 10.1186/s42466-022-00184-x. PMID 35599302